CLINICAL TRIAL: NCT01568099
Title: A Randomized, Controlled, Parallel Group, Patient-blinded, Single-center, Phase I Pilot Study to Assess Tolerability and Safety of Repeated Subcutaneous Administration of Two Doses of AFFITOPE® PD01A Formulated With Adjuvant to Patients With Parkinson's Disease
Brief Title: Tolerability and Safety of Subcutaneous Administration of Two Doses of AFFITOPE® PD01A in Early Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFF008; 2011-002650-31 (EudraCT Number)
Record Dates: First submitted 2012-03-16; First posted 2012-04-02 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: AFFITOPE® PD01A + Adjuvant (Experimental): 4 injections of 15µg AFFITOPE® PD01A/ adjuvanted, once every 4 weeks
  Interventions: Biological: AFFITOPE® PD01A
- B: AFFITOPE® PD01A + Adjuvant (Experimental): 4 injections of 75µg AFFITOPE® PD01A/ adjuvanted, once every 4 weeks
  Interventions: Biological: AFFITOPE® PD01A
- Control (Other): Untreated control group
  Interventions: Other: Control

INTERVENTIONS:
Biological: AFFITOPE® PD01A — s.c. injection
  Arms: A: AFFITOPE® PD01A + Adjuvant; B: AFFITOPE® PD01A + Adjuvant
Other: Control — Untreated control
  Arms: Control

SUMMARY:
This is a phase I study to assess the tolerability and safety of 4 injections of two different doses of AFFITOPE® PD01A formulated with an adjuvant to patients with early Parkinson's disease in male and female patients aged 45 to 65 years (or age between 40 and 45 years if there is no evidence for genetic forms of the disease and the diagnosis of idiopathic Parkinson's disease was confirmed, after approval by Sponsor). One study site in Vienna (Austria) will be involved. Each patient's participation will last 1 year.

In addition, up to 8 patients will be offered participation within an untreated control group.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent capability
* Early PD (≤ 4 years), Hoehn&Yahr Stages I/II and fulfill the UK Parkinson's Disease Society Brain Bank Criteria
* Brain magnetic resonance imaging (MRI) scan and DAT-SPECT scan are consistent with the diagnosis of PD
* Age between 45 and 65 years or age between 40 and 45 years if there is no evidence for genetic forms of the disease and the diagnosis of idiopathic PD was confirmed, after approval by Sponsor
* Caregiver able to attend all visits with patient
* Stable doses of medications (levodopa (+/- benserazide, carbidopa), COMT inhibitors (entacapone, tolcapone), non-ergot dopamine agonists (pramipexol, ropinirol, rotigotine), the MAO-B inhibitor rasagiline and amantadine are allowed)

Exclusion Criteria:

* Women of childbearing potential without birth control or pregnant women
* Participation in another clinical trial
* Autoimmune disease or allergy to components of the vaccine
* Contraindications for MRI, DAT-SPECT, colonoscopy including biopsy or lumbar puncture
* Dementia
* History of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia)
* Active infectious disease
* Immunodeficiency
* Significant systemic illness or psychiatric illness
* Parkinson-like disease secondary to drug therapy side effects
* Parkinson-plus syndromes
* Heredodegenerative disorders
* Alcoholism or substance abuse
* Prior treatment with experimental immunotherapeutics for PD including IVIG, with immunosuppressive drugs or treatment with deep brain stimulation
* Venous status rendering it impossible to place an i.v. access

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tolerability/Safety | 12 month
  * Occurrence of any AE (including a clinical grading scale of AEs according to NCI-CTCAE Version 4.02 (2009) for assessments of AEs + toxicity and including a grading of local injection site reactions according to the FDA Guidance for Industry: Toxicity Scale for Healthy Adult and Adolescents Patients Enrolled in Preventive Vaccine Clinical Trials (2007))
  * Occurrence of any SAE
  * Withdrawal criteria (number of patients who withdraw due to AEs/ reason for withdrawal)

SECONDARY OUTCOMES:
Immunological | 12 month
  - Titer of vaccination induced antibodies directed towards vaccine components, alpha- and beta synuclein
Clinical Activity | 12 month
  * Change in motor symptoms (MDS-UPDRS III)
  * Change in non-motor PD symptoms (e.g.; MDS-UPDRS Ia, II, PDQ39, cognition)
  * Change in biological and radiological markers (e.g. CSF alpha synuclein levels)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Volc, Prim. Dr., Principal Investigator — Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Skodagasse 32, 1080 Vienna
Locations (1):
- Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Skodagasse 32, 1080 Vienna, Vienna, Austria

REFERENCES:
- [Derived] McFarthing K, Simuni T. Clinical Trial Highlights: Targetting Alpha-Synuclein. J Parkinsons Dis. 2019;9(1):5-16. doi: 10.3233/JPD-189004. No abstract available. PMID 30741694